CLINICAL TRIAL: NCT03813238
Title: A Randomized, Double-Blind, Placebo-Controlled Study of TEV-50717 (Deutetrabenazine) for the Treatment of Dyskinesia in Cerebral Palsy in Children and Adolescents
Brief Title: A Study of TEV-50717 (Deutetrabenazine) for the Treatment of Dyskinesia in Cerebral Palsy in Children and Adolescents
Acronym: RECLAIM-DCP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV50717-CNS-30080; 2018-003742-17 (EudraCT Number)
Record Dates: First submitted 2019-01-22; First posted 2019-01-23 (Actual); Results first posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Cerebral Palsy, Dyskinetic
Keywords: DCP
MeSH Terms: conditions — Cerebral Palsy | interventions — deutetrabenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TEV-50717 (Experimental): administered as oral tablets at a starting dose of 6 mg once daily
  Interventions: Drug: TEV-50717
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TEV-50717 — Dosage ranging from 6 mg to 48 mg.
  Other Names: Deutetrabenazine, (previously SD-809)
  Arms: TEV-50717
Drug: Placebo — Dosage ranging from 6 mg to 48 mg.
  Arms: Placebo

SUMMARY:
CP (cerebral palsy) refers to a group of neurological disorders that appear in infancy or early childhood and permanently affect body movement and muscle coordination. CP is caused by damage to or abnormalities inside the developing brain that disrupt the brain's ability to control movement and maintain posture and balance. The signs of CP usually appear in the early months of life, although specific diagnosis may be delayed until the age of 2 years or older. TEV-50717 (deutetrabenazine, also known as SD-809) has already provided evidence for safe and effective use in 2 other hyperkinetic movement disorders, namely chorea in Huntington's disease (HD) and tardive dyskinesia (TD). Currently, there is no approved treatment available for Dyskinesia in cerebral palsy (DCP). The available treatment options address some of the manifestations of DCP. The study population will include pediatric and adolescent participants (6 through 18 years of age) with DCP with predominant choreiform movement disorder, who have had nonprogressive CP symptoms since infancy (≤2 years of age). Diagnosis of DCP is based on the Surveillance of Cerebral Palsy in Europe criteria.

This is a Phase 3 study that will evaluate the efficacy and safety of TEV-50717 administered as oral tablets at a starting dose of 6 mg once daily in participants (age 6 through 18 years, inclusive) with DCP with predominant choreiform movement disorder. The study will be conducted in multiple centers and will use 2 parallel treatment groups (ie, TEV-50717 and placebo) in which participants will be randomized in a 2:1 ratio.

"Predominant" in this instance indicates that the choreiform movement disorder is the main cause of impairment or distress.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 6 through 18 years of age (inclusive) at baseline.
* Participant weighs at least 26 pounds (12 kg) at baseline.
* Participant has had CP symptoms since infancy (≤2 years)
* Choreiform is the prevalent movement disorder as assessed by the EAB at screening.
* Participant has a diagnosis of DCP
* Participant is able to swallow study medication whole.
* Females who are postmenarchal or ≥12 years of age whose male partners are potentially fertile (ie, no vasectomy) must use highly effective birth control methods for the duration of the study
* Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Participant has a predominant movement disorder other than dyskinesia.
* Participant's predominant motor symptoms are dystonic.
* Participant's predominant motor symptoms are spastic.
* Participant has choreiform movement disorder that has not been consistent throughout the life of the participant.
* Participant has clinically significant depression at screening or baseline.
* Note: Participants receiving antidepressant therapy may be enrolled if on a stable dose for at least 6 weeks before screening.
* Participant has a history of suicidal intent or related behaviors within 2 years of screening:
* Previous intent to act on suicidal ideation with a specific plan, irrespective of level of ambivalence, at the time of suicidal thought
* Previous suicidal preparatory acts or behavior
* Participant has a history of a previous actual, interrupted, or aborted suicide attempt.
* Participant has a first-degree relative who has completed suicide.
* Participant has received treatment with stem cells, deep brain stimulation, transmagnetic stimulation, or transcranial direct current stimulation for treatment of abnormal movements or CP within 6 months of the screening visit, or the participant is not in a stable clinical condition.
* Participant has recent surgical procedure or is anticipated to have a surgical procedure during the study that, in the opinion of the investigator, makes the Participant unsuitable for the study.
* Participant has a severe mental disability or an unstable or serious medical illness (eg, epilepsy) at screening or baseline that, in the opinion of the investigator, could jeopardize or would compromise the Participant's ability to participate in this study.
* Participant has a known allergy to any of the components of the investigational medicinal product (IMP).
* Participant is pregnant or breastfeeding.
* Participant has a history of or acknowledges alcohol or substance abuse in the 12 months before screening
* Participants with a history of torsade de pointes, congenital long QT syndrome, bradyarrhythmias, other cardiac arrhythmias, or uncompensated heart failure.
* Additional criteria apply, please contact the investigator for more information

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (70):
- United States (23):
  - Teva Investigational Site 14137, Birmingham, Alabama
  - Teva Investigational Site 14224, Phoenix, Arizona
  - Teva Investigational Site 14227, Loma Linda, California
  - Teva Investigational Site 14295, San Diego, California
  - Teva Investigational Site 14293, Washington D.C., District of Columbia
  - Teva Investigational Site 14127, Miami, Florida
  - Teva Investigational Site 14125, Tampa, Florida
  - Teva Investigational Site 14136, Atlanta, Georgia
  - Teva Investigational Site 14291, Atlanta, Georgia
  - Teva Investigational Site 14130, Savannah, Georgia
  - Teva Investigational Site 14290, New Orleans, Louisiana
  - Teva Investigational Site 14226, Saint Paul, Minnesota
  - Teva Investigational Site 14134, Lincoln, Nebraska
  - Teva Investigational Site 14122, Gibbsboro, New Jersey
  - Teva Investigational Site 14297, New Brunswick, New Jersey
  - Teva Investigational Site 14225, New York, New York
  - Teva Investigational Site 14123, Rochester, New York
  - Teva Investigational Site 14348, Portland, Oregon
  - Teva Investigational Site 14299, Charleston, South Carolina
  - Teva Investigational Site 14129, Nashville, Tennessee
  - Teva Investigational Site 14228, Houston, Texas
  - Teva Investigational Site 14223, Richmond, Virginia
  - Teva Investigational Site 14135, Everett, Washington
- Belgium (2):
  - Teva Investigational Site 37100, Luxembourg City
  - Teva Investigational Site 37102, Woluwe-Saint-Lambert
- Teva Investigational Site 11165, Nepean, Ontario, Canada
- Teva Investigational Site 39058, Copenhagen, Denmark
- Israel (4):
  - Teva Investigational Site 80144, Jerusalem
  - Teva Investigational Site 80145, Safed
  - Teva Investigational Site 80146, Tel Aviv
  - Teva Investigational Site 80147, Ẕerifin
- Italy (6):
  - Teva Investigational Site 30217, Florence
  - Teva Investigational Site 30214, Milan
  - Teva Investigational Site 30213, Napoli
  - Teva Investigational Site 30216, Pisa
  - Teva Investigational Site 30215, Roma
  - Teva Investigational Site 30212, Roma
- Poland (7):
  - Teva Investigational Site 53434, Gdansk
  - Teva Investigational Site 53428, Gdansk
  - Teva Investigational Site 53433, Gmina Strzelin
  - Teva Investigational Site 53427, Krakow
  - Teva Investigational Site 53431, Lublin
  - Teva Investigational Site 53432, Poznan
  - Teva Investigational Site 53430, Wiązowna
- Russia (9):
  - Teva Investigational Site 50477, Kazan'
  - Teva Investigational Site 50475, Khabarovsk
  - Teva Investigational Site 50473, Moscow
  - Teva Investigational Site 50470, Moscow
  - Teva Investigational Site 50485, Nizhny Novgorod
  - Teva Investigational Site 50468, Novosibirsk
  - Teva Investigational Site 50469, Smolensk
  - Teva Investigational Site 50478, Stavropol
  - Teva Investigational Site 50474, Tyumen
- Slovakia (2):
  - Teva Investigational Site 62054, Banská Bystrica
  - Teva Investigational Site 62053, Dubnica nad Váhom
- Spain (6):
  - Teva Investigational Site 31259, Córdoba
  - Teva Investigational Site 31256, Granada
  - Teva Investigational Site 31255, Madrid
  - Teva Investigational Site 31257, Madrid
  - Teva Investigational Site 31258, Seville
  - Teva Investigational Site 31254, Valencia
- Ukraine (5):
  - Teva Investigational Site 58313, Dnipropetrovsk
  - Teva Investigational Site 58312, Kharkiv
  - Teva Investigational Site 58309, Kyiv
  - Teva Investigational Site 58311, Odesa
  - Teva Investigational Site 58310, Vinnytsia
- United Kingdom (4):
  - Teva Investigational Site 34246, Bristol
  - Teva Investigational Site 34245, Edinburgh
  - Teva Investigational Site 34243, London
  - Teva Investigational Site 34244, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo administered as oral tablets once daily for up to 15 weeks.
- TEV-50717: TEV-50717 administered as oral tablets once daily for up to 15 weeks (7 weeks dose titration and 8 weeks maintenance). From Week 1 through Week 7, the dose of TEV-50717 was adjusted according to the titrations scheme (based on body weight and CYP2D6 impairment status at baseline) to identify a dose level that optimally reduced dyskinesia (as determined by the investigator, as indicated by a reduction in the ClinRO of the assessment of the CGI-I) and was well tolerated. After titration, participants continued to receive their maintenance dose over the next 8 weeks.
Period: Overall Study
Arm/Group | Placebo | TEV-50717
Started | 22 | 41
Received at Least 1 Dose of Study Drug | 22 | 40
Modified Intent-to-treat (mITT) Analysis Set (All randomized participants with at least 1 postbaseline centrally read Movement Disorder-Childhood Rating Scale (MD-CRS) part II assessment.) | 21 | 40
Completed | 21 | 30
Not Completed | 1 | 11
Not completed — Adverse Event | 0 | 6
Not completed — Withdrawal by parent/guardian | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other than specified | 1 | 2

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TEV-50717 | Total
Number analyzed (Participants) | 22 | 41 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.5 (3.98) | 11.3 (3.14) | 11.3 (3.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 12 | 29 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 20 | 36 | 56
  Unknown or Not Reported | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 21 | 40 | 61
  Race: Other | 1 | 1 | 2
MD-CRS Part II Total Score (Movement Disorder Severity, Centrally Read) [Mean (Standard Deviation); unit: units on a scale] — MD-CRS part II evaluates the severity of movement disorder in a scale of 0 to 4 in 7 body regions, where 0 = absence of a movement disorder and 4 = movement disorder is present during all tasks for the region examined and/or involves 3 or more of other regions. The 7 body regions are eye and periorbital region, face, tongue and perioral region, neck, trunk, upper limb, and lower limb. Total score was obtained by summing the individual items scores and ranges from 0 (absent of a movement disorder) to 28 (marked/prolonged movement disorder), with higher scores indicating more movement disorder. Population: The mITT analysis set included all randomized participants with at least 1 postbaseline centrally read MD-CRS part II assessment.
  units on a scale
    number analyzed (Participants) | 21 | 40 | 61
    (all) | 10.4 (6.09) | 11.7 (6.85) | 11.3 (6.58)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Movement Disorder-Childhood Rating Scale (MD-CRS) Part II Total Score (Movement Disorder Severity, Centrally Read) at Week 15
Description: MD-CRS part II evaluates the severity of movement disorder in a scale of 0 to 4 in 7 body regions, all areas in which dyskinesia can be seen. All items were scored by the rater in the clinic and were centrally read based on video recording. In rating the movement disorder of body part, 0 refers to absence of a movement disorder and 4 refers to a situation where movement disorder is present during all of the tasks for the region examined and/or involves 3 or more of the other regions, making completion impossible. The 7 body regions are (i) eye and periorbital region, (ii) face, (iii) tongue and perioral region, (iv) neck, (v) trunk, (vi) upper limb, and (vii) lower limb. Total score was obtained by summing the individual items scores and ranges from 0 (absent of a movement disorder) to 28 (marked/prolonged movement disorder), with higher scores indicating more movement disorder. Least square (LS) mean and standard error (SE) was calculated using a mixed-model repeated-measures (MMRM).
Time Frame: Baseline, Week 15
Population: The mITT analysis set included all randomized participants with at least 1 postbaseline centrally read MD-CRS part II assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 21 | 40
units on a scale | -0.4 (1.09) | -1.5 (0.88)
Statistical Analysis 1: Comparison: Placebo vs TEV-50717; The LS mean of the change in MDCRS part II total score from baseline to Week 15 was compared (TEV-50717 arm versus placebo) using a 1-sided test for superiority at a nominal significance level of α=0.025; Test type: Superiority; p = 0.335, Mixed Models Analysis; LS mean difference = -1.2, 95% CI 2-sided [-3.49 to 1.19]

2. Secondary Outcome: Change From Baseline in the MD-CRS Part I Total Score (General Assessment, Centrally Read) at Week 15
Description: The MD-CRS part I evaluates the impact of dyskinesia in cerebral palsy (DCP) on the activities of the participant and provides a general assessment of the movement disorder of motor function (7 items), oral/verbal function (3 items), self-care (3 items), and attention/alertness (2 items) on a scale of 0 (present) to 4 (absent). All items were scored by the rater in the clinic and were centrally read based on video recording. The total score was obtained by summing the individual items scores and ranges from 0 (marked/prolonged disorder) to 60 (absent of a disorder), with higher scores indicating lesser disorder.
Time Frame: Baseline, Week 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 21 | 40
units on a scale | -0.8 (2.51) | -0.7 (2.10)

3. Secondary Outcome: Caregiver Global Impression of Improvement (CaGI-I) Scale Score (Global, Caregiver Rated) at Week 15
Description: The CaGI-I is single item questionnaire to assess the caregiver's impression of improvement in dyskinesia symptoms after initiating therapy. The scale is a caregiver-reported outcome that aims to evaluate all aspects of participants' health and determine if there has been an overall improvement or not in dyskinesia symptoms. The caregiver selected the 1 response from the response options that gave the most accurate description of change in dyskinesia symptoms of the participant they cared for from the beginning of the study: 1=very much improved (since the initiation of treatment); 2=much improved; 3=minimally improved; 4=no change from baseline (symptoms remain essentially unchanged); 5=minimally worse; 6=much worse; 7=very much worse (since the initiation of treatment).
Time Frame: Week 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 21 | 40
units on a scale | 3.3 (0.83) | 3.3 (0.84)

4. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) Scale Score (Global, Physician Rated) at Week 15
Description: CGI-I is a clinician-reported outcome that uses a 7-point Likert scale that allows the clinician to compare participant's condition at the visit to the baseline condition as follows: 1=very much improved since initiation of treatment (nearly all better; good level of functioning; minimal symptoms; represents a very substantial change); 2=much improved (notably better with significant reduction of symptoms; increase in the level of functioning but some symptoms remain); 3=minimally improved (slightly better with little or no clinically meaningful reduction of symptoms; represents very little change in basic clinical status, level of care, or functional capacity); 4=no change from baseline (symptoms remain unchanged); 5=minimally worse (slightly worse but may not be clinically meaningful); 6=much worse (clinically significant increase in symptoms and diminished functioning); 7=very much worse since the initiation of treatment (severe exacerbation of symptoms and loss of functioning).
Time Frame: Week 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 21 | 40
units on a scale | 3.5 (0.87) | 3.4 (0.78)

5. Secondary Outcome: Change From Baseline in Unified Huntington's Disease Rating Scale-Total Maximal Chorea (UHDRS-TMC) Score (Centrally Read) at Week 15
Description: The UHDRS-TMC is part of the Unified Huntington's Disease Rating Scale-Total Motor Score (UHDRS-TMS) assessment and assesses the severity of chorea in the 7 body parts: face, mouth, trunk, and the 4 extremities (right and left upper extremities, right and left lower extremities). Each part was rated from 0 (absent) to 4 (prolonged). The central rating was done for all participants, based on the videos collected for the central rating of MD-CRS. The TMC score was obtained by adding up each of the separate scores and ranged from 0 (absent) to 28 (marked/prolonged), with higher scores indicating the worse symptoms.
Time Frame: Baseline, Week 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 21 | 40
units on a scale | 0.3 (2.87) | -1.2 (2.52)

6. Secondary Outcome: Change From Baseline in Unified Huntington's Disease Rating Scale-Total Maximal Dystonia (UHDRS-TMD) Score (Centrally Read) at Week 15
Description: The UHDRS-TMD is part of the UHDRS-TMS assessment and assesses the severity of dystonia in the 5 body parts: trunk and the 4 extremities (right and left upper extremities, right and left lower extremities). Each part was rated from 0 (absent) to 4 (prolonged). The central rating was done for all participants, based on the videos collected for the central rating of MD-CRS. The TMD score was obtained by adding up each of the separate scores and ranged from 0 (absent) to 20 (marked/prolonged), with higher scores indicating the worse symptoms.
Time Frame: Baseline, Week 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 21 | 40
units on a scale | -0.6 (1.46) | -0.2 (1.19)

7. Secondary Outcome: Change From Baseline in the MD-CRS Part I Total Score (General Assessment, Physician Rated) at Week 15
Description: The MD-CRS part I evaluates the impact of DCP on the activities of the participant and provides a general assessment of the movement disorder of motor function (7 items), oral/verbal function (3 items), self-care (3 items), and attention/alertness (2 items) on a scale of 0 (present) to 4 (absent). All items were scored by the investigational center physician. The total score was obtained by summing the individual items scores and ranges from 0 (marked/prolonged movement disorder) to 60 (absent of a movement disorder), with higher scores indicating lesser movement disorder.
Time Frame: Baseline, Week 15
Population: The mITT analysis set included all randomized participants with at least 1 postbaseline centrally read MD-CRS part II assessment. Here, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 21 | 31
units on a scale | -0.7 (3.21) | -1.0 (3.57)

8. Secondary Outcome: Change From Baseline in the MD-CRS Part II Total Score (General Assessment, Physician Rated) at Week 15
Description: The MD-CRS part II evaluates the severity of the movement disorder in a scale of 0 to 4 in 7 body regions, all areas in which dyskinesia can be seen in participants with CP. All items were scored by the investigational center physician. In rating the movement disorder of the body part, 0 refers to absence of a movement disorder and 4 refers to a situation where movement disorder is present during all of the tasks for the region examined and/or involves 3 or more of the other regions, making completion impossible. The 7 body regions are (i) eye and periorbital region, (ii) face, (iii) tongue and perioral region, (iv) neck, (v) trunk, (vi) upper limb, and (vii) lower limb. The total score was obtained by summing the individual items scores and ranges from 0 (absent of a movement disorder) to 28 (marked/prolonged movement disorder), with higher scores indicating more movement disorder.
Time Frame: Baseline, Week 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 21 | 31
units on a scale | -1.5 (3.20) | -2.4 (3.15)

9. Secondary Outcome: Change From Baseline in MD-CRS Global Index Score (Calculated From MD-CRS Parts I and II Total Scores, Physician Rated) at Week 15
Description: The MD-CRS Global Index is a global measure of the MD-CRS that consolidates the information from parts I and II using the method of weighted means of the 2 normalized indexes obtained from each part. The standardized/normalized score for each item of MD-CRS parts I and II with value X is calculated using the formula: Xst = X - Xmin divided by Xmax - Xmin, where Xmax is the maximum value for the score, and Xmin is the minimum value for the score, or 4 and 0 respectively. The normalized index for the scale, MD-CRS parts I or II, Index I or II, is calculated as the mean value of Xst. The MD-CRS Global Index is the weighted mean of the normalized indexes for centrally read MD-CRS parts I and II using the formula: Global index = n1 * index 1 + n2 * index 2 divided by n1 + n2, where n1 and n2 are the numbers of items in MD-CRS parts I and II respectively. The minimum score is 0 (better) and the maximum score is 1 (worse). The higher score indicates more severe movement disorder.
Time Frame: Baseline, Week 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 21 | 31
units on a scale | -0.0 (0.06) | -0.0 (0.06)

10. Secondary Outcome: Change From Baseline in MD-CRS Global Index Score (Calculated From MD-CRS Parts I and II Total Scores, Centrally Read) at Week 15
Description: as for outcome 9
Time Frame: Baseline, Week 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 21 | 31
units on a scale | -0.0 (0.08) | -0.0 (0.06)

11. Secondary Outcome: Change From Baseline in UHDRS-TMS Score (Physician Rated) at Week 15
Description: The UHDRS comprises a broad assessment of features associated with Huntington's disease (HD). It is a research tool that has been developed to provide a uniform assessment of the clinical features and course of HD. The Total Motor Score assessment of the UHDRS (UHDRS-TMS) comprises 15 items and assesses eye movements, speech, alternating hand movements, dystonia, chorea, and gait. The UHDRS-TMS was calculated as the sum of the 31 motor assessments; each of which ranged between 0 (absent) to 4 (worst). All items were scored by the investigational center physician. TMS score is a sum of individual scores ranging from 0 (normal motor function) to 124 (severely impaired motor function), with lower scores indicating better motor function.
Time Frame: Baseline, Week 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 21 | 31
units on a scale | -4.1 (8.35) | -7.6 (10.28)

12. Secondary Outcome: Change From Baseline in UHDRS-TMC Score (Physician Rated) at Week 15
Description: The UHDRS-TMC is part of the UHDRS-TMS assessment and assesses the severity of chorea in the 7 body parts: face, mouth, trunk, and the 4 extremities (right and left upper extremities, right and left lower extremities). Each part was rated from 0 (absent) to 4 (prolonged). All items were scored by the investigational center physician. The TMC score was obtained by adding up each of the separate scores and ranged from 0 (absent) to 28 (marked/prolonged), with higher scores indicating the worse symptoms.
Time Frame: Baseline, Week 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 21 | 31
units on a scale | -2.2 (4.05) | -2.9 (3.50)

13. Secondary Outcome: Change From Baseline in UHDRS-TMD Score (Physician Rated) at Week 15
Description: The UHDRS-TMD is part of the UHDRS-TMS assessment and assesses the severity of dystonia in the 5 body parts: trunk and the 4 extremities (right and left upper extremities, right and left lower extremities). Each part was rated from 0 (absent) to 4 (prolonged). All items were scored by the investigational center physician. The TMD score was obtained by adding up each of the separate scores and ranged from 0 (absent) to 20 (marked/prolonged), with higher scores indicating the worse symptoms.
Time Frame: Baseline, Week 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 21 | 31
units on a scale | 0.6 (1.86) | -1.3 (1.56)

14. Secondary Outcome: Change From Baseline in Pediatric Evaluation Disability Inventory-Computer Adapted Test (PEDI-CAT) Score (Activities of Daily Living [ADL], Caregiver Completed, Content-Balanced Version) at Week 15
Description: The PEDI-CAT measures function in 4 domains: (1) Daily Activities; (2) Mobility; (3) Social/Cognitive, and (4) Responsibility. The content balanced version presents a balance of items from each of the Daily Activities domain's content areas (Getting Dressed, Keeping Clean, Home Tasks, and Eating and Mealtime). A total of approximately 30 items were administered. PEDI-CAT software utilizes Item Response Theory statistical models to estimate a child's abilities from a minimal number of the most relevant items or from a set number of items within each domain. The CAT program then displays the results: normative standard scores, scaled scores and SE. Scaled score is reported in this endpoint. Scaled scores are based on an estimate of the placement of an individual child along the hierarchical scale within each domain. PEDI-CAT scaled scores are currently on a 20 (lesser improvement) to 80 (more improvement) scale metric. Higher scores indicate greater improvement in functional skills.
Time Frame: Baseline, Week 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 16 | 29
units on a scale | -0.4 (1.78) | -0.6 (3.22)

15. Secondary Outcome: Change From Baseline in the CP Module of the Pediatric Quality of Life Inventory (PedsQL) Total Score (Quality of Life [QoL], Participant/Caregiver) at Week 15
Description: The 35-item PedsQL 3.0 CP module encompasses 7 scales: Daily Activities (9 items); School Activities (4 items); Movement and Balance (5 items); Pain and Hurt (4 items); Fatigue (4 items); Eating Activities (5 items); and Speech and Communication (4 items). For children ages 6 and 7 years and 8 to 12 years, a child self-report and a parent proxy report are completed. For children ages 13 to 18 years, no parent proxy report is required. A 5-point response scale is utilized across child self-report and parent proxy report: 0=never a problem; 1=almost never a problem; 2=sometimes a problem; 3=often a problem; 4=almost always a problem. Items are reverse scored and linearly transformed to a 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0), so that higher scores indicate better quality of life (fewer problems). Total score was computed as the sum of 35 items divided by the number of items answered. Change from baseline scores can range from -100 to 100.
Time Frame: Baseline, Week 15
Population: The mITT analysis set included all randomized participants with at least 1 postbaseline centrally read MD-CRS part II assessment. Here, overall number of participants analyzed = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable for specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 18 | 33
units on a scale
  Self-report | 1.9 (11.17) | 3.2 (14.96)
  Proxy-report: number analyzed (Participants) | 11 | 23
  Proxy-report | 4.1 (8.80) | -0.7 (16.46)

16. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Scale Score (Global, Participant/Caregiver) at Week 15
Description: The PGI-I is single item questionnaire to assess the participant's impression of improvement in dyskinesia symptoms after initiating therapy. The scale is a participant-reported outcome that aims to evaluate all aspects of participants' health and determine if there has been an overall improvement or not in dyskinesia symptoms. The participant selected the 1 response from the visual response options ("emojis") that gave the most accurate description of his/her state of health and overall status: 1=much improved (since the initiation of treatment); 2=somewhat improved; 3=no change; 4=somewhat worse; 5=much worse (since the initiation of treatment).
Time Frame: Week 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 20 | 31
units on a scale | 2.4 (0.81) | 2.4 (0.80)

17. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S) Scale Score (Global, Physician Rated) at Week 15
Description: The CGI-S uses a 7-point Likert scale to assess dyskinesia severity as follows (with anchor points for choosing the most appropriate severity level caused by DCP): 1=normal (not at all ill, symptoms of disorder not present past 7 days); 2=borderline (subtle or suspected pathology); 3=mild (clearly established symptoms with minimal, if any, distress or difficulty in social and/or occupational function); 4=moderate (overt symptoms causing noticeable, but modest, functional impairment or distress; symptom level may warrant medication); 5=marked (intrusive symptoms that distinctly impair social/occupational function or cause intrusive levels of distress); 6=severe (disruptive symptoms, behavior and function are frequently influenced by symptoms, may require assistance from others); 7=extreme (symptoms drastically interferes in many life functions; may be hospitalized).
Time Frame: Baseline, Week 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 21 | 31
units on a scale | -0.6 (0.75) | -0.7 (0.78)

18. Secondary Outcome: Number of Participants With CaGI-I Response
Description: CaGI-I response was defined as participants who were described by the caregiver as "Much Improved" or "Very Much Improved" in the CaGI-I score. The CaGI-I is single item questionnaire to assess the caregiver's impression of improvement in dyskinesia symptoms after initiating therapy. The scale is a caregiver-reported outcome that aims to evaluate all aspects of participants' health and determine if there has been an overall improvement or not in dyskinesia symptoms. The caregiver selected the 1 response from the response options that gave the most accurate description of change in dyskinesia symptoms of the participant they cared for from the beginning of the study: 1=very much improved (since the initiation of treatment); 2=much improved; 3=minimally improved; 4=no change from baseline (symptoms remain essentially unchanged); 5=minimally worse; 6=much worse; 7=very much worse (since the initiation of treatment).
Time Frame: Week 15
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 20 | 31
Participants | 4 | 8

19. Secondary Outcome: Number of Participants With CGI-I Response
Description: CGI-I response was defined as participants who were described as "Much Improved" or "Very Much Improved" in the CGI-I score. CGI-I is a clinician-reported outcome that uses a 7-point Likert scale that allows the clinician to compare participant's condition at the visit to the baseline condition as follows: 1=very much improved since initiation of treatment (nearly all better; good level of functioning; minimal symptoms); 2=much improved (notably better with significant reduction of symptoms; increase in the level of functioning but some symptoms remain); 3=minimally improved (slightly better with little or no clinically meaningful reduction of symptoms); 4=no change from baseline (symptoms remain unchanged); 5=minimally worse (slightly worse but may not be clinically meaningful); 6=much worse (clinically significant increase in symptoms and diminished functioning); 7=very much worse since the initiation of treatment (severe exacerbation of symptoms and loss of functioning).
Time Frame: Week 15
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 21 | 31
Participants | 4 | 6

20. Secondary Outcome: Number of Participants With CGI-S Response
Description: CGI-S response was defined as participants who had a reduction of ≥1 point in the CGI-S score. The CGI-S uses a 7-point Likert scale to assess dyskinesia severity as follows (with anchor points for choosing the most appropriate severity level caused by DCP): 1=normal (not at all ill, symptoms of disorder not present past 7 days); 2=borderline (subtle or suspected pathology); 3=mild (clearly established symptoms with minimal, if any, distress or difficulty in social and/or occupational function); 4=moderate (overt symptoms causing noticeable, but modest, functional impairment or distress; symptom level may warrant medication); 5=marked (intrusive symptoms that distinctly impair social/occupational function or cause intrusive levels of distress); 6=severe (disruptive symptoms, behavior and function are frequently influenced by symptoms, may require assistance from others); 7=extreme (symptoms drastically interferes in many life functions; may be hospitalized).
Time Frame: Week 15
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 21 | 31
Participants | 9 | 17

21. Secondary Outcome: Number of Participants With PGI-I Response
Description: PGI-I response was defined as participants who were described as "Much Improved" or "Somewhat Improved" in the PGI-I score. The PGI-I is single item questionnaire to assess the participant's impression of improvement in dyskinesia symptoms after initiating therapy. The scale is a participant-reported outcome that aims to evaluate all aspects of participants' health and determine if there has been an overall improvement or not in dyskinesia symptoms. The participant selected the 1 response from the visual response options ("emojis") that gave the most accurate description of his/her state of health and overall status: 1=much improved (since the initiation of treatment); 2=somewhat improved; 3=no change; 4=somewhat worse; 5=much worse (since the initiation of treatment).
Time Frame: Week 15
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 20 | 31
Participants | 9 | 18

22. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. SAEs included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'.
Time Frame: Baseline up to Week 17
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 22 | 40
Participants | 15 | 35

23. Secondary Outcome: Number of Participants With Shift From Baseline to Week 15 in Electrocardiogram (ECG) Findings
Description: The number of participants with a difference (shift) from baseline in any of the following ECG parameters is reported by group: Heart rate, PR interval, QRS interval, RR interval, QT interval, and QT interval corrected using the Fridericia formula (QTcF). Shifts represented as Baseline - Week 15 value (last observed postbaseline value).
Time Frame: Baseline to Week 15
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug. Here, overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 20 | 32
Participants
  Normal - Normal | 14 | 20
  Normal - Abnormal | 1 | 5
  Abnormal - Normal | 1 | 3
  Abnormal - Abnormal | 4 | 4

24. Secondary Outcome: Change From Baseline in Child Behavior Checklist (CBCL) Competence Total Score at Week 15
Description: The CBCL assesses behavioral and emotional status in children ages 6 through 18 years of age as reported by the caregiver. The full CBCL has two parts, a Competence Scale (Parts I to VII) and a Syndrome Scale (behavioral items). The Competence Scale (Parts I to VII) assesses various activities (for example, sports, hobbies, games, organizations, clubs, teams, groups, jobs, and chores), interpersonal relationships, and academic performance. The checklists having 120 questions consist of a number of statements about the child's behavior and responses which are recorded on a scale: 0 = Not True; 1 = Somewhat or Sometimes True; 2 = Very True or Often True. CBCL competence total score ranged from 0 (no problem) to 240 (lesser problem), was calculated by adding individual score of each domain. Higher scores indicate greater problems in child behavior.
Time Frame: Baseline, Week 15
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 12 | 28
units on a scale | -1.12 (4.279) | -0.08 (2.716)

25. Secondary Outcome: Change From Baseline in Child Behavior Checklist (CBCL) Syndrome Total Score at Week 15
Description: The CBCL assesses behavioral and emotional status in children ages 6 through 18 years of age as reported by the caregiver. The full CBCL has two parts, a Competence Scale (Parts I to VII) and a Syndrome Scale (behavioral items). The Syndrome Scale comprises 113 questions related to problem behaviors. For each item, the responses are recorded on a scale: 0 = Not True; 1 = Somewhat or Sometimes True; 2 = Very True or Often True. The problem behaviors are scored on the following 8 empirically based syndromes: anxious/depressed, withdrawn/depressed, somatic complaints, social problems, thought problems, attention problems, rule-breaking behavior, and aggressive behavior. CBCL syndrome total score ranged from 0 (no problem) to 226 (lesser problem), was calculated by adding individual score of each domain. Higher scores indicate greater problems in child behavior.
Time Frame: Baseline, Week 15
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 20 | 31
units on a scale | -7.1 (11.34) | -11.6 (15.23)

26. Secondary Outcome: Change From Baseline in Extrapyramidal Symptom Rating Scale (ESRS) Subscale I Total Score at Week 15
Description: The ESRS subscale I is a 7-item subjective questionnaire to evaluate parkinsonism, akathisia, dystonia and dyskinesia. The ESRS I is scored on 4-point scale (0=absent, 1=Mild, 2=Moderate, 3=Severe) for each item. The evaluation takes into account the verbal report of the participant on 1) the frequency and duration of the symptom during the day, 2) the number of days the symptom was present during the last week, and 3) the subjective evaluation of the intensity of the symptom by the participant. Total score was the sum of the 7 items which ranges from 0 (absent) to 28 (severe). Higher scores indicate greater severity of disorder.
Time Frame: Baseline, Week 15
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 21 | 31
units on a scale | -1.4 (1.40) | -1.5 (2.08)

27. Secondary Outcome: Change From Baseline in Extrapyramidal Symptom Rating Scale (ESRS) Subscale II Total Score at Week 15
Description: The ESRS subscale II is a 17-item questionnaire to evaluate parkinsonism and akathisia. The ESRS II consists of the following parts: tremor (0 [none]-48 [severe]), gait and posture (0 [none]-6 [severe]), postural stability (0 [none]-6 [severe]), rigidity (0 [none]-24 [severe]), expressive automatic movements (0 [none]-6 [severe]), bradykinesia (0 [none]-6 [severe]), and akathisia (0 [none]-6 [severe]). Total score was the sum of the 17 items which from ranges from 0 (absent) to 102 (severe). Higher scores indicate greater severity of disorder.
Time Frame: Baseline, Week 15
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 21 | 31
units on a scale | -2.6 (5.64) | -1.8 (6.37)

28. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) Total Score at Week 15
Description: The ESS is a self-administered questionnaire composed of 8 questions that provide a measure of a participant's general level of daytime sleepiness. The ESS is composed of 8 items. The responders were asked to rate their chances of falling asleep while engaged at 8 different activities, on a 4-point scale: 0 = would never fall asleep; 1=slight chance of falling asleep; 2=moderate chance of falling asleep; 3=high chance of falling asleep. Total score was calculated as the sum of 8 item scores which ranges from 0 (never) to 24 (high chance of falling asleep). Higher scores indicate high chances of falling asleep.
Time Frame: Baseline, Week 15
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 20 | 29
units on a scale | -0.9 (1.74) | 1.6 (5.21)

29. Secondary Outcome: Number of Participants With Columbia-Suicide Severity Rating Scale (C-SSRS) Outcomes (Suicidal Ideation and Suicidal Behavior) at Week 15
Description: Participants were placed into categories for suicidal ideation and suicidal behavior based on their responses to various questions. For suicidal ideation, following categories were used: None; Wish to be dead; Non-specific active suicidal thoughts; Any methods (not plan) without intent to act; Some intent to act, without specific plan; and Specific plan and intent. For suicidal behavior, following categories were used: None; Preparatory acts or behavior; Aborted attempt; Interrupted attempt; Actual attempt; and Suicide. Number of participants with suicidal ideation and/or suicidal behavior at Week 15 are reported.
Time Frame: Week 15
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TEV-50717
Number analyzed (Participants) | 8 | 9
Participants
  Suicidal ideation - None | 8 | 9
  Suicidal ideation - Wish to be dead | 0 | 0
  Suicidal ideation - Non-specific active suicidal thoughts | 0 | 0
  Suicidal ideation - Any methods (not plan) without intent to act | 0 | 0
  Suicidal ideation - Some intent to act, without specific plan | 0 | 0
  Suicidal ideation - Specific plan and intent | 0 | 0
  Suicidal behavior - None | 8 | 9
  Suicidal behavior - Preparatory acts or behavior | 0 | 0
  Suicidal behavior - Aborted attempt | 0 | 0
  Suicidal behavior - Interrupted attempt | 0 | 0
  Suicidal behavior - Actual attempt | 0 | 0
  Suicidal behavior - Suicide | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 17
Description: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Placebo | TEV-50717
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/40
Other Adverse Events (participants affected / at risk) | 10/22 | 34/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | TEV-50717 (N=40)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (6)
Fatigue (General disorders) | 0 (0) | 4 (5)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (3) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Weight increased (Investigations) | 0 (0) | 3 (3)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Drooling (Nervous system disorders) | 1 (1) | 4 (4)
Dysarthria (Nervous system disorders) | 0 (0) | 2 (2)
Dyskinesia (Nervous system disorders) | 0 (0) | 2 (2)
Dystonia (Nervous system disorders) | 1 (1) | 4 (5)
Lethargy (Nervous system disorders) | 0 (0) | 2 (3)
Somnolence (Nervous system disorders) | 0 (0) | 17 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT03813238/Prot_002.pdf
  • Statistical Analysis Plan (2022-05-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT03813238/SAP_003.pdf